CLINICAL TRIAL: NCT03817437
Title: Correlation Study Between Socio-economical Deprivation and Oral Health in in French Children of 9 Years of Age in 2017. A Nationwide Database Retrospective Observational Cohort Study
Brief Title: Correlation Study Between Socio-economical Deprivation and Oral Health in Children of 9 Years of Age
Acronym: PRECA-6
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0401
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Tooth Decay; Missing Tooth/Teeth
Keywords: Oral health; Odontology; Epidemiology; Public health; Deprivation
MeSH Terms: conditions — Dental Caries; Anodontia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective, observational cohort study.

Objectives :

To search for correlations between socio-economical deprivation and oral health in french children of 9 years of age.

To study the annual use of oral and dental care of children from 6 to 9 years of age depending on their geographical and socio-economical environment, and the medical demography ; To identify and study the share of the cohort not using oral and dental care, and the socio-economical and geographical factors implicated in this non-use of care.

The study will use data from the french nationwide healthcare systems database (SNDS) and data from the french national institute of statistics and economic studies (INSEE).

ELIGIBILITY:
Inclusion criteria:

* Being born in 2008
* Being covered by the mandatory french national health insurance plan without discontinuity between 2014 and 2017
* Living in France without discontinuity between 2014 and 2017

Exclusion criteria:

- None

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients born in 2008
Sampling Method: Non-Probability Sample
Enrollment: 600000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Correlations (odds-ratios) between several socio-economical indicators and oral care use | 36 months
  Correlations (odds-ratios) between several socio-economical indicators and oral care use

SECONDARY OUTCOMES:
Mean numbers of several types of oral cares depending on the patients geographical and socio-economical environment | 36 months
  Mean numbers of several types of oral cares depending on the patients geographical and socio-economical environment, and the medical demography

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BOUREL, MsC, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC